CLINICAL TRIAL: NCT05141019
Title: Trial of Preemptive Pharmacogenetics in Underserved Patients
Acronym: ToPP-UP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB202101316 -N; R01HG011800 (NIH)
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Use of Prescription Medications; Pharmacogenetic Testing
Keywords: Pharmacogenetics; Medically underserved; Implementation; Effectiveness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate panel-based pharmacogenetic genotyping (Experimental): Subjects assigned to the immediate pharmacogenetic genotyping group will be tested and have their results both entered into their electronic health record as well as provided to them within 2-4 weeks from enrollment.
  Interventions: Diagnostic Test: Panel-based pharmacogenetic genotyping
- Delayed panel-based pharmacogenetic genotyping (Other): Subjects assigned to delayed panel-based pharmacogenetic genotyping will be tested, but their results will not be released until after their participation in the study has ended (12 months after enrollment).
  Interventions: Diagnostic Test: Panel-based pharmacogenetic genotyping

INTERVENTIONS:
Diagnostic Test: Panel-based pharmacogenetic genotyping — After providing consent, subjects will be randomized to receive either the immediate pharmacogenetic testing arm or the delayed arm. Subjects in both groups will provide a DNA sample by saliva, buccal cell, or blood at study enrollment. Subjects assigned to the immediate pharmacogenetic genotyping group will be tested and will have their results entered into their electronic health record (EHR) and provided to them within 2-4 weeks. Subjects assigned to the delayed pharmacogenetic genotyping group will also be tested, but their results will not be released until after their participation in the study has ended. Subjects in each arm will complete surveys and questionnaires regarding their medication satisfaction, as well as their healthcare utilization use at baseline and then again at 6- and 12-months. Implementation-specific questions will also be asked to assess the feasibility and sustainability of the intervention as well as assessments of intervention fidelity and adaptations.

SUMMARY:
This proposed research is relevant to human health because preemptive clinical pharmacogenetic testing may improve the personalization of drug therapy which should improve patient outcomes. Better understanding of the effectiveness and feasibility of preemptive clinical pharmacogenetic testing will inform when and how this innovative healthcare technology is implemented into clinical care. To ensure equitable dissemination in all patient populations, such data is also needed in racial minorities and other traditionally underserved populations. The combined proposed research are relevant to the parts of the NIH's mission pertaining to protecting and improving health and developing scientific human resources that will ensure the Nation's capability to prevent and treat disease.

DETAILED DESCRIPTION:
Preemptive pharmacogenetic (PGx) testing may be particularly beneficial in medically underserved populations by reducing the number of appointments required to optimize drug therapy and increasing the effectiveness of less expensive off-patent medications - the type most often with pharmacogenetic guidelines available (PGx drugs). However, there is little data available to guide clinical implementation in these patient populations. Our long-term goal is to contribute toward the efficient implementation of PGx into clinical practice to improve the precision of medication prescribing. The overall objective for this application is to identify PGx drug usage patterns in medically underserved patients, and assess the feasibility and effectiveness of preemptive PGx testing in this patient population. The central hypothesis is that medically underserved patients are prescribed more PGx drugs, and preemptive PGx testing is feasible as well as effective in improving patient medication satisfaction. The rationale for the proposed research is that identifying patient populations that can most benefit from PGx testing will facilitate clinical implementation that may reduce medication treatment disparities.

The investigators plan to test the central hypothesis and accomplish the overall objective of this application by pursuing three specific aims. The first aim is to identify clinical, demographic and socioeconomic factors associated with PGx drug prescribing patterns in a large, real-world, diverse patient population. The investigators will accomplish this aim by comparing clinical, demographic, and socioeconomic data with prescription data from millions of patients across the State of Florida. The second aim is to develop a low-cost, ancestrally inclusive PGx testing panel designed to inform commonly used PGx drugs. The investigators will design a low-cost, clinically validated panel that will include variants common in racial minorities in the U.S. The investigators plan to leverage extensive batching of tests and an already available genotyping platform that minimizes labor costs in order to achieve significant cost savings. The third aim is to determine the feasibility of low-cost preemptive PGx testing in a medically underserved population as well as its effect on patient medication satisfaction. The investigators will accomplish this aim by completing a randomized open-label clinical trial comparing medically underserved patients receiving preemptive PGx testing to those receiving usual care. The investigators will compare key implementation metrics and will also conduct semi-structured interviews in both patients and healthcare providers to assess PGx perceptions of feasibility and sustainability from stakeholders.

The proposed research is significant because it should contribute valuable preliminary data toward both the real-world effectiveness of preemptive PGx testing as well as the feasibility of studying and implementing this technology in medically underserved patients - an area of PGx research where few data are available. The proposed research is innovative because this project will utilize additional demographic and socioeconomic data that, with along with clinical data, should better identify patient populations most likely to benefit from PGx testing and allow focused of implementation efforts to those populations. Ultimately, the investigators expect to have developed valuable data identifying patients most likely to benefit from preemptive PGx testing, particularly in patients who are medically underserved and/or members of racial minorities. These results should have an important positive impact because they can inform further clinical implementation efforts of PGx as well as future large clinical trials of preemptive testing, ideally reducing healthcare disparities in the field of precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years of age
* at least 3 active prescriptions documented within medical records
* Experienced a change to an active prescription within the past 8 months, defined by:
* Addition of a new medication
* Change in the dose of a current medication
* Diagnosis of any condition that could be treated with a medication that can be informed by the pharmacogenetic testing panel.

This will likely include:

* generalized depression or anxiety disorder
* gastroesophageal reflux disorder
* erosive esophagitis
* gastric ulcer
* acute coronary syndrome
* chronic pain
* surgery (orthopedic, gastrointestinal, cardiovascular etc.)
* osteoarthritis
* Dyslipidemia
* Heart failure
* Deep vein thrombosis
* Atrial fibrillation
* Moderate to severe trauma
* stroke
* hypercholesterolemia
* conditions requiring chronic anticoagulation

Exclusion Criteria:

* Any history of previous pharmacogenetic testing
* Any medical condition that would prohibit the ability to answer study questions
* History of Allogenic stem cell or liver transplant
* History of chronic kidney dialysis
* Life expectancy less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Treatment Satisfaction Measured by the Treatment Satisfaction Questionnaire for Medication (TSQM) | 12-14 months
  The primary feasibility outcome will be change in patient treatment satisfaction between baseline and 12 months after enrollment into the study. This patient-reported outcome will be measured via the TSQM. The TSQM is a validated tool that assesses three medication-related domains (effectiveness, side effects, and convenience) to synthesize a global satisfaction score. Both global satisfaction and scores from individual domains will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Duarte, PharmD, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT05141019/ICF_001.pdf